CLINICAL TRIAL: NCT02571530
Title: Phase 1 Trial of Super-selective Intra-arterial Cerebral Infusion of Trastuzumab After Blood-Brain Barrier Disruption for the Treatment of Cerebral Metastases of HER2/Neu Positive Breast Cancer
Brief Title: Super-selective Intra-arterial Cerebral Infusion of Trastuzumab for the Treatment of Cerebral Metastases of HER2/Neu Positive Breast Cancer
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Northwell Health (Other)
Responsible Party: Principal Investigator, John Boockvar, MD Zucker SOM @Hofstra/Northwell, Professor, Northwell Health
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 15-312
Record Dates: First submitted 2015-09-16; First posted 2015-10-08 (Estimated); Last update posted 2021-11-03 (Actual); Status verified 2021-10

CONDITIONS: Neoplasm Metastasis
MeSH Terms: conditions — Neoplasm Metastasis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Intra-arterial Cerebral Infusion of Trastuzumab (Experimental): Super-selective Intra-arterial Cerebral Infusion of Trastuzumab After Blood-Brain Barrier Disruption
  Interventions: Drug: Intra-arterial Cerebral Infusion of Trastuzumab

INTERVENTIONS:
Drug: Intra-arterial Cerebral Infusion of Trastuzumab

SUMMARY:
The purpose of this study is to evaluate the safety of administering a single dose of trastuzumab into the artery for the treatment of brain metastasis(es) from HER2/neu positive breast cancer.

This study will try to determine the best tolerated single dosage of trastuzumab administered into arteries by gradually increasing the dosage given to participants as the study progresses. Early participants will receive a dosage of 1 mg/kg. As more participants enroll into the study, this single dosage will be increased at designated levels up to 8 mg/kg, if it's determined to be safe to increase.

Trastuzumab is a type of antibody, which is a protein used by the body's immune system to fight against pathogens such as bacteria and viruses. This antibody binds to cell receptors known as the HER2/neu tyrosine kinase receptor. These receptors are expressed in certain cancer subtypes such as breast cancer. By blocking signaling through this HER2/neu receptor, trastuzumab can slow down or stop the over-expression of the HER2/neu protein. Over-expression of HER2/neu has been shown to play a role in the development and progression of certain types of breast cancer. Therefore, by slowing down or stopping the expression of HER2/neu, investigators hope to slow down or stop the growth of metastasis(es) and increase the responsiveness to therapy.

ELIGIBILITY:
Inclusion Criteria:

1. Male and female patients 18 years of age or older
2. Karnofsky Performance Status (KPS) of 70 or higher
3. Capable of giving informed consent or have an acceptable surrogate capable of giving consent of the subject's behalf
4. Have a documented history of HER2/neu positive breast cancer that is 3+ on immunohistochemical staining or positive on fluorescent in-situ hybridization (FISH) or chromogenic in-situ hybridization (CISH) and have evidence of parenchymal metastatic tumor(s) on brain imaging studies.
5. Adequate labs for procedure with trastuzumab, including but not limited to White Blood Count (WBC), Hemoglobin, Hematocrit, Platelet Count, Prothrombin Time (PT), International Normalized Ratio (INR), Sodium, Potassium, Chloride, Glucose, Blood Urea Nitrogen (BUN), Serum Creatinine (CR)

Exclusion Criteria:

1. Age less than 18 years
2. KPS less than 70
3. Brain metastases without history of HER2/neu positive breast cancer
4. Leptomeningeal dissemination of brain metastases
5. Pregnancy or refusal to use contraception during a 3 month period before and 7 month period after Intra-arterial (IA) trastuzumab administration
6. Prior administration of intraarterial trastuzumab
7. Subjects with inadequate baseline Left Ventricular Ejection Fraction (LVEF)
8. Subjects with history of infusion reaction with trastuzumab
9. Subjects who have had blood brain barrier (BBB) disruption with mannitol within 48 hours
10. Subjects with evidence of midline shift or herniation
11. Subjects with resectable brain metastases or whose cerebral tumors are amenable to stereotactic radio-surgery
12. Subjects who have not progressed after therapy for brain metastases

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2 (Actual)
Dates: Start 2015-08 (Actual); Primary Completion 2021-06 (Actual); Study Completion 2021-06 (Actual)

PRIMARY OUTCOMES:
Maximum tolerated dose (MTD) | 30 days
  Maximum tolerated dose (MTD) the highest dose at which there are no dose limiting toxicities.
Adverse events and dose-limiting toxicities | 30 days
  A dose-limiting toxicity (DLT) will be defined as any grade 3 or 4 NCI Common Toxicity Criteria adverse event (CTCAE V4.0).

SECONDARY OUTCOMES:
Response Evaluation Criteria in Solid Tumors (RECIST) | 1 year
  RECIST Criteria
Overall Survival (OS) | 1 year
Intracranial Time to Progression | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Lenox Hill Brain Tumor Center, New York, New York, United States